CLINICAL TRIAL: NCT06492564
Title: An Exploratory Study to Establish the Dose, Safety and Pathogenicity of a SARS-CoV-2 Omicron Challenge Strain (BA.5) in Healthy Participants 18 to 40 Years of Age
Brief Title: Dose, Safety and Pathogenicity of SARS-CoV-2 (COVID-19) Omicron Virus (BA.5)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HRD-vCS-003
Record Dates: First submitted 2024-07-05; First posted 2024-07-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Omicron; COVID-19; Human Challenge Trials
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): Low dose, expected to be approximately 10^4 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Interventions: Biological: SARS-CoV-2 omicron virus dose arm 1
- Dose 2 (Experimental): Medium dose, expected to be approximately 10^5 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Interventions: Biological: SARS-CoV-2 omicron virus dose arm 2
- Dose 3 (Experimental): High dose, expected to be approximately 10^6 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Interventions: Biological: SARS-CoV-2 omicron virus dose arm 3

INTERVENTIONS:
Biological: SARS-CoV-2 omicron virus dose arm 1 — Low dose, approximately 10^4 TCID50/mL
  Arms: Dose 1
Biological: SARS-CoV-2 omicron virus dose arm 2 — Medium dose, approximately 10^5 TCID50/mL
  Arms: Dose 2
Biological: SARS-CoV-2 omicron virus dose arm 3 — High dose, approximately 10^6 TCID50/mL
  Arms: Dose 3

SUMMARY:
An Exploratory Study to Establish the Dose, Safety and Pathogenicity of a SARS-CoV-2 Omicron Challenge Strain (BA.5) in Healthy Participants 18 to 40 Years of Age

DETAILED DESCRIPTION:
This is an exploratory study of an SARS-CoV-2 Omicron (BA.5) challenge strain to determine the optimum safe infectious titer of challenge agent in healthy participants 18 to 40 years of age.

Up to 90 participants who meet all study inclusion and no exclusion criteria will be allocated to one of the three dose escalating cohorts (Dose 1, Dose 2 or Dose 3), with up to 30 participants in each dose group, to receive one dose of SARS-CoV-2 omicron. Based on the outcome of each cohort the next cohort may receive a high or lower dose than the previous cohort.

Each participant will remain in the study for approximately 9 months from screening to the last clinic visit.

The study is divided into three phases:

1. Screening phase: Screening will occur between Day -90 to Day -2/-1.
2. Quarantine phase: Participants will stay in the quarantine unit for approximately 17 days (from Day -2/-1 to Day 14).

   One or two days prior to the day of inoculation with the challenge virus, participants will be admitted to quarantine where their eligibility will be reassessed. If participants remain eligible for the study, they will receive the challenge virus on Day 0. Participants will undergo a range of clinical assessments and safety monitoring for the entirety of their stay in quarantine. Participants will be discharged from the quarantine unit on Day 14 (or may remain longer at the principal investigator's discretion). If participants do not become infected with the virus they may be discharged earlier on Day 8.
3. Outpatient phase:Following the conclusion of the quarantine phase, participants will receive telephone follow up calls every 3 days between quarantine discharge and the day 28 follow up visit. Participants will also attend additional Follow-Up visits, approximately 28 days, 90 days, and 180 days after they received the study virus. Their symptoms will be reassessed, and a complete safety examination performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult male or female aged between 18 and 40 years
* A total body weight ≥50 kg and body mass index (BMI) ≥18 kg/m2 and ≤28kg/m2. The upper limit of BMI may be increased to ≤30kg/m2 at the PI's discretion, in the case of physically fit muscular individuals.
* In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety.
* Documented medical history
* Adherence to contraception requirements
* Serosuitable for the challenge virus
* Participants must have been previously vaccinated with a COVID-19 vaccine licensed for use in the UK and completed the course

Exclusion Criteria:

* History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit.
* Any history or evidence of any clinically significant or currently active disease.
* Any participants who have smoked ≥5 pack years at any time.
* Female participants who are breastfeeding, or have been pregnant within 6 months prior to the study, or have a positive pregnancy test at any point during screening or prior to inoculation.
* Any history of anaphylaxis and/or a any history of severe allergic reaction.
* Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
* History of severe COVID-19 or severe complication of any other viral disease.
* Participants with no knowledge of their family history, as deemed appropriate by the PI
* Significant abnormality of the nose, includes loss of or alterations in smell or taste,nasal polyps, epistaxis, nasal or sinus surgery.
* Recent vaccinations or intention to receive vaccination before the Day 28 follow up visit. Receipt of COVID-19 vaccine in the last 3 months prior to inoculation and/or a diagnosis of COVID 19 confirmed by a physician within the last 6 months prior to screening or at any time between screening and quarantine admission.
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned inoculation or planned during the 3 months after the final visit.
* Recent receipt of investigational drugs or challenge viruses.
* Use or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows.
* Positive drugs of abuse test or recent history or presence of alcohol addiction
* A forced expiratory volume in 1 second (FEV1) <80%.
* Positive HIV, hepatitis B virus, or hepatitis C virus test.
* Presence of fever, defined as participant presenting with a temperature reading of ≥37.9°C on Day -2/-1 and/or pre-inoculation on Day 0.
* Those employed or immediate relatives of those employed at hVIVO or the sponsor.
* Any other reason, in the opinion of the investigator deems the participant unsuitable for the study
* Sensitivity to any of the study interventions, challenge agent or components thereof (including lactose), or drug or other allergy that, in the opinion of the PI/investigator, contraindicates participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events related to the viral challenge | Day 0 to Day 28
  Number of participants with challenge Agent-emergent adverse events (AEs) at least possibly related to the viral challenge from viral challenge (Day 0) up to the Day 28 follow-up
Occurrence of Serious Adverse Events and Medically Attended Adverse Events, related to the viral challenge | Day 0 to Day 180
  Occurrence of serious AEs (SAEs) and Medically Attended Adverse Events (MAAEs) related to the viral challenge from viral challenge (Day 0) up to the Day 180 follow-up
Induces laboratory-confirmed infection in ≥40% of inoculated participants | Day 1 to Day 14
  Quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR)-confirmed SARS-CoV-2 omicron infection, defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (reported over 4 planned consecutive assessments within 48 hours), from Day 1 pm to planned discharge from quarantine (Day 14 am).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bevan, MBBS, Principal Investigator — hVIVO Services Ltd.
Locations (1):
- hVIVO Services Ltd, 40 Bank Street, Canary Wharf, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No